CLINICAL TRIAL: NCT02131064
Title: A Randomized, Multicenter, Open-Label, Two-Arm, Phase III Neoadjuvant Study Evaluating Trastuzumab Emtansine Plus Pertuzumab Compared With Chemotherapy Plus Trastuzumab and Pertuzumab for Patients With HER2-Positive Breast Cancer
Brief Title: A Study Evaluating Trastuzumab Emtansine Plus Pertuzumab Compared With Chemotherapy Plus Trastuzumab and Pertuzumab for Participants With Human Epidermal Growth Factor Receptor 2 (HER2)-Positive Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO28408; TRIO021 (Other: Roche); 2012-004879-38 (EudraCT Number)
Record Dates: First submitted 2014-05-02; First posted 2014-05-06 (Estimated); Results first posted 2017-06-08 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Carboplatin; Docetaxel; pertuzumab; Trastuzumab; Ado-Trastuzumab Emtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trastuzumab (TCH) + Pertuzumab (Active Comparator): Participants will receive pertuzumab 840 milligrams (mg) (loading dose) and 420 mg (maintenance dose) intravenous (IV) infusion followed by trastuzumab 8 milligrams per kilogram (mg/kg) (loading dose) and 6 mg/kg (maintenance dose) IV infusion followed by docetaxel 75 milligrams per square meter (mg/m^2) IV infusion and carboplatin at a dose to achieve an area under the curve (AUC) of 6 milligrams per milliliter* minute (mg/mL*min) IV infusion every 3 weeks (q3w) for 6 cycles in neoadjuvant period. Participants will receive pertuzumab 840 mg (loading dose) and 420 mg (maintenance dose) IV infusion followed by trastuzumab 8 mg/kg (loading dose) and 6 mg/kg (maintenance dose) IV infusion q3w for rest of the cycles (12 cycles) in adjuvant period (up to a total of 18 cycles).
  Interventions: Drug: Carboplatin; Drug: Docetaxel; Drug: Pertuzumab; Drug: Trastuzumab
- Trastuzumab Emtansine (T-DM1) + Pertuzumab (Experimental): Participants will receive pertuzumab 840 mg (loading dose) and 420 mg (maintenance dose) IV infusion followed by trastuzumab emtansine 3.6 mg/kg IV infusion q3w for a total of 18 cycles (6 cycles of neoadjuvant period and 12 cycles of adjuvant period).
  Interventions: Drug: Pertuzumab; Drug: Trastuzumab Emtansine

INTERVENTIONS:
Drug: Carboplatin — Carboplatin IV infusion at a dose to achieve an AUC of 6 mg*min/mL q3w
  Arms: Trastuzumab (TCH) + Pertuzumab
Drug: Docetaxel — Docetaxel 75 mg/m^2 IV infusion q3w
  Arms: Trastuzumab (TCH) + Pertuzumab
Drug: Pertuzumab — Pertuzumab 840 mg (loading dose); and 420 mg (maintenance dose) IV infusion q3w
  Other Names: Perjeta®, RO4368451
Drug: Trastuzumab — Trastuzumab 8 mg/kg (loading dose); and 6 mg/kg (maintenance dose) IV infusion q3w
  Other Names: Herceptin®
  Arms: Trastuzumab (TCH) + Pertuzumab
Drug: Trastuzumab Emtansine — Trastuzumab Emtansine 3.6 mg/kg IV infusion q3w
  Other Names: Kadcyla®, RO5304020
  Arms: Trastuzumab Emtansine (T-DM1) + Pertuzumab

SUMMARY:
This is a randomized, multicenter, open-label, two-arm study in treatment-naive participants with operable, locally advanced, or inflammatory, centrally-assessed HER2-positive early breast cancer (EBC) whose primary tumors were greater than or equal to (>/=) 2 centimeters (cm). The study was designed to evaluate the efficacy and safety of trastuzumab emtansine + pertuzumab (experimental arm; T-DM1 + P) versus chemotherapy, trastuzumab + pertuzumab (control arm; TCH + P). The study comprised a neoadjuvant treatment period, followed by surgery, and an adjuvant treatment period.

Treatment can be stopped due to disease recurrence, unacceptable toxicity, withdrawal of consent, or study termination.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive breast cancer with a primary tumor size of greater than (>) 2 cm
* HER2-positive breast cancer
* Participants with multifocal tumors (more than one tumor confined to the same quadrant as the primary tumor) are eligible provided all discrete lesions are sampled and centrally confirmed as HER2 positive
* Stage at presentation: cT2-cT4, cN0-cN3, cM0, according to American Joint Committee on Cancer (AJCC) staging system
* Known hormone receptor status of the primary tumor
* Participant agreement to undergo mastectomy or breast-conserving surgery after neoadjuvant therapy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Baseline Left Ventricular Ejection Fraction (LVEF) >/= 55 percent (%) measured by echocardiogram (ECHO) or multiple-gated acquisition (MUGA)
* Effective contraception as defined by protocol

Exclusion Criteria:

* Stage IV (metastatic) breast cancer
* Participants who have received prior anti-cancer therapy for breast cancer except those participants with a history of breast lobular carcinoma in situ (LCIS) that was surgically managed or ductal carcinoma in situ (DCIS) treated exclusively with mastectomy. In case of prior history of LCIS/DCIS, >5 years must have passed from surgery until diagnosis of current breast cancer
* Participants with multicentric (multiple tumors involving more than 1 quadrant) or bilateral breast cancer
* Participants who have undergone incisional and/or excisional biopsy of primary tumor and/or axillary lymph nodes
* Axillary lymph node dissection or positive sentinel lymph node prior to start of neoadjuvant therapy
* History of concurrent or previously non-breast malignancies except for appropriately treated (1) non-melanoma skin cancer and (2) in situ carcinomas, including cervix, colon, and skin. A participant with previous invasive non-breast cancer is eligible provided he/she has been disease-free >/= 5 years
* Treatment with any investigational drug within 28 days prior to randomization
* Current National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version (v) 4.0
* Any significant concurrent medical or surgical conditions or findings that would jeopardize the participant's safety or ability to complete the study
* Current pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 444 (Actual)
Dates: Start 2014-06-25 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2018-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (79):
- United States (16):
  - St. Jude Heritage Healthcare; Virgiia K.Crosson Can Ctr, Fullerton, California
  - Cancer Care Assoc Med Group, Los Angeles, California
  - Coastal Integrative Cancer Care, San Luis Obispo, California
  - Central Coast Medical Oncology, Santa Maria, California
  - UCLA Hematology/Oncology, Santa Monica, California
  - Memorial Cancer Institute, Hollywood, Florida
  - Md Anderson Cancer Center Orlando, Orlando, Florida
  - New England Cancer Specialists, Scarborough, Maine
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - ProHEALTH Care Associates LLP, Lake Success, New York
  - Montefiore Medical Center, The Bronx, New York
  - Hope A Women's Cancer Center, Asheville, North Carolina
  - Levine Cancer Institute, Charlotte, North Carolina
  - Roper Bon Secours St. Francis Cancer Center, Charleston, South Carolina
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
- Belgium (5):
  - UZ Antwerpen, Edegem
  - UZ Leuven Gasthuisberg, Leuven
  - Clinique Saint-Joseph, Liège
  - Clinique Ste-Elisabeth, Pharmacie, Namur
  - Sint Augustinus Wilrijk, Wilrijk
- Canada (6):
  - Cross Cancer Institute ; Dept of Medical Oncology, Edmonton, Alberta
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael'S Hospital, Toronto, Ontario
  - Chum Hospital Notre Dame, Montreal, Quebec
  - McGill University; Sir Mortimer B Davis Jewish General Hospital; Oncology, Montreal, Quebec
  - CHU de Québec - Hôpital du Saint-Sacrement / ONCOLOGY, Québec
- France (9):
  - Ico - Paul Papin, Angers
  - HOPITAL JEAN MINJOZ; Oncologie, Besançon
  - Hopital Morvan, Brest
  - CHD Les Oudairies, La Roche-sur-Yon
  - Centre Oscar Lambret, Lille
  - Institut Paoli Calmettes, Marseille
  - Centre Catherine De Sienne, Nantes
  - Centre Rene Gauducheau, Saint-Herblain
  - Nouvel Hopital Civil - CHU Strasbourg, Strasbourg
- Germany (5):
  - Klinikum Sindelfingen-Böblingen; Frauenklinik, Böblingen
  - Luisenkrankenhaus GmbH, Brustzentrum, Düsseldorf
  - Universitätsklinikum Erlangen; Frauenklinik, Erlangen
  - Universitätsklinikum Mainz, Mainz
  - Interdisziplinäres Onkologisches Zentrum, München
- Russia (6):
  - Moscow City Oncology Hospital #62, Moscovskaya Oblast, Moscow Oblast
  - Regional Oncology Hospital Of Kursk; Chemotherapy, Kislino, Kursk Region
  - S.I. Russian Oncological Research Center n.a. N.N. Blokhin, Moscow
  - State Inst. Of Healthcare Orenburg Regional Clinical Oncology Dis, Orenburg
  - Saint-Petersburg City Clinical Oncology Dispensary, Saint Petersburg
  - Railway Clinical Hospital on Saratov - 2 Station Oao "Rzhd", Saratov
- South Korea (6):
  - National Cancer Center, Gyeonggi-do
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Asan Medical Center - Oncology, Seoul
  - Samsung Medical Center, Seoul
- Spain (16):
  - Corporacio Sanitaria Parc Tauli; Servicio de Oncologia, Sabadell, Barcelona
  - IInstituto Oncologico de San Sebastian, Oncologikoa; Servicio de Oncologia, Donostia / San Sebastian, Guipuzcoa
  - Hospital Universitari de Lleida Arnau de Vilanova, Lleida, Lerida
  - Complejo Hospitalario Universitario A Coruña (CHUAC, Materno Infantil), Oncología, A Coruña
  - Hospital Nuestra Señora de Sonsoles; servicio de Oncologia, Ávila
  - Hospital del Mar; Servicio de Oncologia, Barcelona
  - Fundacio Santa Creu I Sant Pau, Barcelona
  - Complejo Hospitalario de Jaen, Jaén
  - Hospital General Universitario Gregorio Marañon; Servicio de Oncologia, Madrid
  - Hospital Universitario Clínico San Carlos; Servicio de Oncologia, Madrid
  - Centro Integral Oncologico Clara Campal (CIOCC); Dirección Médica, Madrid
  - Hospital Quiron de Madrid; Servicio de Oncologia, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Universitario Miguel Servet; Servicio Oncologia, Zaragoza
- Taiwan (6):
  - Kaohsiung Medical Uni Chung-Ho Hospital; Dept of Surgery, Kaohsiung City
  - National Taiwan Uni Hospital, Taipei
  - Mackay Memorial Hospital; Dept of Surgery, Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center; Hemato-Oncology, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
- Ukraine (4):
  - Cherkassy Regional Oncological Hospital, Cherkassy
  - State Medical Academy; Oncology, Dnipropetrovsk
  - Karkiv Regional Oncology Center, Kharkiv
  - Lvov State Regional Center, Lviv

REFERENCES:
- [Derived] de Haas SL, Slamon DJ, Martin M, Press MF, Lewis GD, Lambertini C, Prat A, Lopez-Valverde V, Boulet T, Hurvitz SA. Tumor biomarkers and efficacy in patients treated with trastuzumab emtansine + pertuzumab versus standard of care in HER2-positive early breast cancer: an open-label, phase III study (KRISTINE). Breast Cancer Res. 2023 Jan 11;25(1):2. doi: 10.1186/s13058-022-01587-z. PMID 36631725
- [Derived] Hurvitz SA, Martin M, Jung KH, Huang CS, Harbeck N, Valero V, Stroyakovskiy D, Wildiers H, Campone M, Boileau JF, Fasching PA, Afenjar K, Spera G, Lopez-Valverde V, Song C, Trask P, Boulet T, Sparano JA, Symmans WF, Thompson AM, Slamon D. Neoadjuvant Trastuzumab Emtansine and Pertuzumab in Human Epidermal Growth Factor Receptor 2-Positive Breast Cancer: Three-Year Outcomes From the Phase III KRISTINE Study. J Clin Oncol. 2019 Sep 1;37(25):2206-2216. doi: 10.1200/JCO.19.00882. Epub 2019 Jun 3. PMID 31157583
- [Derived] Hurvitz SA, Martin M, Symmans WF, Jung KH, Huang CS, Thompson AM, Harbeck N, Valero V, Stroyakovskiy D, Wildiers H, Campone M, Boileau JF, Beckmann MW, Afenjar K, Fresco R, Helms HJ, Xu J, Lin YG, Sparano J, Slamon D. Neoadjuvant trastuzumab, pertuzumab, and chemotherapy versus trastuzumab emtansine plus pertuzumab in patients with HER2-positive breast cancer (KRISTINE): a randomised, open-label, multicentre, phase 3 trial. Lancet Oncol. 2018 Jan;19(1):115-126. doi: 10.1016/S1470-2045(17)30716-7. Epub 2017 Nov 23. PMID 29175149

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 574 participants were screened at 65 sites in 10 countries, of which 444 participants were randomized in two arms: Trastuzumab (TCH) + Pertuzumab (P) (Arm A) and Trastuzumab Emtansine (TDM1) + P (Arm B)
Groups:
- TCH + P: Participants received pertuzumab 840 milligrams (mg) (loading dose) and 420 mg (maintenance dose) intravenous (IV) infusion, trastuzumab 8 milligrams per kilogram (mg/kg) (loading dose) and 6 mg/kg (maintenance dose) IV infusion, docetaxel 75 milligrams per square meter (mg/m^2) IV infusion and carboplatin at a dose to achieve an area under the curve (AUC) of 6 milligrams per milliliter* minute (mg/mL*min) IV infusion every 3 weeks (q3w) for 6 cycles in neoadjuvant period. Participants received pertuzumab 840 mg (loading dose) and 420 mg (maintenance dose) IV infusion followed by trastuzumab 8 mg/kg (loading dose) and 6 mg/kg (maintenance dose) IV infusion q3w for rest of the cycles (12 cycles) in adjuvant period (up to a total of 18 cycles).
- T-DM1 + P: Participants received pertuzumab 840 mg (loading dose) and 420 mg (maintenance dose) IV infusion followed by trastuzumab emtansine 3.6 mg/kg IV infusion q3w for a total of 18 cycles (6 cycles of neoadjuvant period and 12 cycles of adjuvant period).
Period: Overall Study
Arm/Group | TCH + P | T-DM1 + P
Started | 221 | 223
Completed | 196 | 189
Not Completed | 25 | 34
Not completed — Death | 5 | 6
Not completed — Lost to Follow-up | 4 | 8
Not completed — Withdrawal by Subject | 14 | 18
Not completed — Other | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TCH + P | T-DM1 + P | Total
Number analyzed (Participants) | 221 | 223 | 444
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.3 (11.2) | 50.5 (10.6) | 49.9 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 221 | 222 | 443
  Male | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Total Pathological Complete Response (tpCR) Assessed Based on Tumor Samples
Description: tpCR was assessed by local pathology review on samples taken at surgery following completion of neoadjuvant therapy. tpCR was defined as the absence of any residual invasive cancer on hematoxylin and eosin evaluation of the resected breast specimen and all sampled ipsilateral lymph nodes ( that is [i.e.], ypT0/is, ypN0 in the American Joint Committee on Cancer [AJCC] staging system, 7th edition). Percentage of participants with tpCR was reported.
Time Frame: Pre-surgery (within 6 weeks after neoadjuvant therapy; up to approximately 6 months)
Population: The Intent-to-treat (ITT) Population comprised all randomized patients, whether or not they received any study treatment or completed a full course of study treatment. Patients were analyzed according to their randomized treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | TCH + P | T-DM1 + P
Number analyzed (Participants) | 221 | 223
Percentage of Participants | 56.1 [49.29 to 62.76] | 44.4 [37.76 to 51.18]
Statistical Analysis 1: Comparison: TCH + P vs T-DM1 + P; 95% CI for the difference in tPCR rates between treatment arms was calculated using normal approximation; Test type: Superiority; p = 0.0126, Cochran-Mantel-Haenszel Chi-Square — Threshold for significance at 5%; The Cochran-Mantel-Haenszel Chi-square test was used and stratified by local hormone receptor status and clinical stage at presentation; Difference in tpCR rate = -11.71, 95% CI 2-sided [-20.95 to -2.48]

2. Secondary Outcome: Overall Survival
Description: Overall survival in the overall study population was defined as the time from the date of randomization to the date of death from any cause. 3 years OS event-free rate per randomized treatment arms in the ITT population were estimated using the Kaplan-Meier method and estimated the probability of a patient being event-free after 3 years after treatment.
Time Frame: From randomization until death (up to approximately 47 months)
Population: The ITT Population comprised all randomized patients, whether or not they received any study treatment or completed a full course of study treatment. Patients were analyzed according to their randomized treatment.
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | TCH + P | T-DM1 + P
Number analyzed (Participants) | 221 | 223
Probability | 97.6 [95.5 to 99.7] | 97.0 [94.6 to 99.4]
Statistical Analysis 1: Comparison: TCH + P vs T-DM1 + P; Test type: Superiority; p = 0.7557, Cochran-Mantel-Haenszel Chi-Square Test; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.21, 95% CI 2-sided [0.37 to 3.96]

3. Secondary Outcome: Percentage of Participants Who Received Breast-Conserving Surgery (BCS)
Description: BCS rate was defined as the percentage of participants who achieve BCS out of the ITT population of participants without inflammatory breast cancer.
Time Frame: Surgery performed after completion of neoadjuvant therapy (approximately 6 months after neoadjuvant period)
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | TCH + P | T-DM1 + P
Number analyzed (Participants) | 213 | 218
Percentage of Participants | 52.6 (45.65) [45.65 to 59.45] | 41.7 (35.12) [35.12 to 48.33]
Statistical Analysis 1: Comparison: TCH + P vs T-DM1 + P; 95% CI for the difference in BCS rate between treatment arms was calculated using normal approximation; Test type: Superiority; p = 0.0228, Cochran-Mantel-Haenszel Chi-Square; [statistical method as in outcome 1, analysis 1]; Difference in BCS rate = -10.84, 95% CI 2-sided [-20.21 to -1.47]

4. Secondary Outcome: Event-Free Survival
Description: Event-free survival (EFS) is defined as the time from randomization to disease progression or disease recurrence (local, regional, distant, or contralateral, invasive or non-invasive), or death from any cause. 3 years EFS rate per randomized treatment arms in the ITT population were estimated using the Kaplan-Meier method and estimated the probability of a patient being event-free after 3 years after treatment.
Time Frame: From randomization up to disease progression or recurrence or death (up to approximately 47 months)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | TCH + P | T-DM1 + P
Number analyzed (Participants) | 221 | 223
Probability | 94.21 [91.02 to 97.39] | 85.28 [80.47 to 90.08]
Statistical Analysis 1: Comparison: TCH + P vs T-DM1 + P; Test type: Superiority; p = 0.0027, Log Rank; The Log Rank was used and stratified by local hormone receptor status and clinical stage at presentation; Hazard Ratio (HR) = 2.61, 95% CI 2-sided [1.36 to 4.98]

5. Secondary Outcome: Invasive Disease-free Survival (IDFS)
Description: IDFS is defined only for participants who undergo surgery. IDFS is defined as the time from surgery to the first documented occurrence of an IDFS event, defined as: Ipsilateral invasive breast tumor recurrence; Ipsilateral local-regional invasive breast cancer recurrence; Distant recurrence; Contralateral invasive breast cancer; and death from any cause. 3 years of IDFS event-free rate per randomized treatment arms in the ITT population were estimated using the Kaplan-Meier method and estimated the probability of a patient being event-free after 3 years after treatment.
Time Frame: From surgery to the first documented occurrence of IDFC event (up to approximately 47 months)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | TCH + P | T-DM1 + P
Number analyzed (Participants) | 221 | 223
Probability | 91.99 [86.73 to 97.26] | 93.04 [89.39 to 96.69]
Statistical Analysis 1: Comparison: TCH + P vs T-DM1 + P; Test type: Superiority; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.52 to 2.40]

6. Secondary Outcome: Percentage of Participants by Response for Neuropathy Single Item
Description: Participants answered the question "Did you have tingling hands/feet?", from the Modified Quality of Life Questionnaire Breast Cancer 23 (mQLQ-BR23), on a 5-point scale (1 'Not at all', 2 'A little', 3 'Somewhat', 4 'Quite a bit', 5 'Very much'). Percentage of participants by each response was reported.
Time Frame: Baseline,Cycle(C) 3,C5 of neoadjuvant period (each C=21 days); pre-surgery visit (within 6weeks after neoadjuvant therapy; up to approx 6months), C4 & 8 of Adjuvant Period (each C=21 days), End of Treatment, Follow up 2 & 4 (approx 47 months)
Population: ITT population of patients with both a baseline assessment and at least one post-treatment assessment in the respective single question are included in the analysis.
Measure: Number; unit: Percentage of Participants
Arm/Group | TCH + P | T-DM1 + P
Number analyzed (Participants) | 221 | 223
Percentage of Participants
  Not at all: Baseline: number analyzed (Participants) | 198 | 204
  Not at all: Baseline | 78.7 | 81.2
  A little bit: Baseline: number analyzed (Participants) | 198 | 204
  A little bit: Baseline | 9.5 | 9.4
  Somewhat: Baseline: number analyzed (Participants) | 198 | 204
  Somewhat: Baseline | 0 | 0
  Quite a bit: Baseline: number analyzed (Participants) | 198 | 204
  Quite a bit: Baseline | 0.9 | 0.9
  Very much: Baseline: number analyzed (Participants) | 198 | 204
  Very much: Baseline | 0.5 | 0
  Not at all: Neoadjuvant Cycle 3: number analyzed (Participants) | 177 | 183
  Not at all: Neoadjuvant Cycle 3 | 54.3 | 59.6
  A little bit: Neoadjuvant Cycle 3: number analyzed (Participants) | 177 | 183
  A little bit: Neoadjuvant Cycle 3 | 20.8 | 19.3
  Somewhat: Neoadjuvant Cycle 3: number analyzed (Participants) | 177 | 183
  Somewhat: Neoadjuvant Cycle 3 | 0 | 0
  Quite a bit: Neoadjuvant Cycle 3: number analyzed (Participants) | 177 | 183
  Quite a bit: Neoadjuvant Cycle 3 | 3.2 | 2.7
  Very much: Neoadjuvant Cycle 3: number analyzed (Participants) | 177 | 183
  Very much: Neoadjuvant Cycle 3 | 1.8 | 0.4
  Not at all: Neoadjuvant Cycle 5: number analyzed (Participants) | 182 | 178
  Not at all: Neoadjuvant Cycle 5 | 37.1 | 54.3
  A little bit: Neoadjuvant Cycle 5: number analyzed (Participants) | 182 | 178
  A little bit: Neoadjuvant Cycle 5 | 29.9 | 21.1
  Somewhat: Neoadjuvant Cycle 5: number analyzed (Participants) | 182 | 178
  Somewhat: Neoadjuvant Cycle 5 | 0 | 0
  Quite a bit: Neoadjuvant Cycle 5: number analyzed (Participants) | 182 | 178
  Quite a bit: Neoadjuvant Cycle 5 | 8.6 | 2.7
  Very much: Neoadjuvant Cycle 5: number analyzed (Participants) | 182 | 178
  Very much: Neoadjuvant Cycle 5 | 6.8 | 1.8
  Not at all: Pre-Surgery: number analyzed (Participants) | 170 | 171
  Not at all: Pre-Surgery | 22.6 | 52.0
  A little bit: Pre-Surgery: number analyzed (Participants) | 170 | 171
  A little bit: Pre-Surgery | 29.0 | 17.9
  Somewhat: Pre-Surgery: number analyzed (Participants) | 170 | 171
  Somewhat: Pre-Surgery | 0 | 0
  Quite a bit: Pre-Surgery: number analyzed (Participants) | 170 | 171
  Quite a bit: Pre-Surgery | 15.4 | 5.4
  Very much: Pre-Surgery: number analyzed (Participants) | 170 | 171
  Very much: Pre-Surgery | 10.0 | 1.3
  Not at all: Adjuvant Cycle 4: number analyzed (Participants) | 174 | 155
  Not at all: Adjuvant Cycle 4 | 31.2 | 42.6
  A little bit: Adjuvant Cycle 4: number analyzed (Participants) | 174 | 155
  A little bit: Adjuvant Cycle 4 | 31.7 | 15.2
  Somewhat: Adjuvant Cycle 4: number analyzed (Participants) | 174 | 155
  Somewhat: Adjuvant Cycle 4 | 0 | 0
  Quite a bit: Adjuvant Cycle 4: number analyzed (Participants) | 174 | 155
  Quite a bit: Adjuvant Cycle 4 | 9.5 | 9.0
  Very much: Adjuvant Cycle 4: number analyzed (Participants) | 174 | 155
  Very much: Adjuvant Cycle 4 | 6.3 | 2.7
  Not at all: Adjuvant Cycle 8: number analyzed (Participants) | 168 | 143
  Not at all: Adjuvant Cycle 8 | 33.0 | 31.8
  A little bit: Adjuvant Cycle 8: number analyzed (Participants) | 168 | 143
  A little bit: Adjuvant Cycle 8 | 28.1 | 19.3
  Somewhat: Adjuvant Cycle 8: number analyzed (Participants) | 168 | 143
  Somewhat: Adjuvant Cycle 8 | 0 | 0
  Quite a bit: Adjuvant Cycle 8: number analyzed (Participants) | 168 | 143
  Quite a bit: Adjuvant Cycle 8 | 10.9 | 9.0
  Very much: Adjuvant Cycle 8: number analyzed (Participants) | 168 | 143
  Very much: Adjuvant Cycle 8 | 4.1 | 4.0
  Not at all: End of Therapy: number analyzed (Participants) | 172 | 165
  Not at all: End of Therapy | 31.2 | 31.4
  A little bit: End of Therapy: number analyzed (Participants) | 172 | 165
  A little bit: End of Therapy | 30.8 | 23.8
  Somewhat: End of Therapy: number analyzed (Participants) | 172 | 165
  Somewhat: End of Therapy | 0 | 0
  Quite a bit: End of Therapy: number analyzed (Participants) | 172 | 165
  Quite a bit: End of Therapy | 10.9 | 12.1
  Very much: End of Therapy: number analyzed (Participants) | 172 | 165
  Very much: End of Therapy | 5.0 | 6.7
  Not at all: Follow-up 2: number analyzed (Participants) | 150 | 136
  Not at all: Follow-up 2 | 38.0 | 32.7
  A little bit: Follow-up 2: number analyzed (Participants) | 150 | 136
  A little bit: Follow-up 2 | 19.9 | 19.3
  Somewhat: Follow-up 2: number analyzed (Participants) | 150 | 136
  Somewhat: Follow-up 2 | 0 | 0
  Quite a bit: Follow-up 2: number analyzed (Participants) | 150 | 136
  Quite a bit: Follow-up 2 | 5.9 | 7.6
  Very much: Follow-up 2: number analyzed (Participants) | 150 | 136
  Very much: Follow-up 2 | 4.1 | 1.3
  Not at all: Follow-up 4: number analyzed (Participants) | 136 | 124
  Not at all: Follow-up 4 | 39.8 | 32.7
  A little bit: Follow-up 4: number analyzed (Participants) | 136 | 124
  A little bit: Follow-up 4 | 15.4 | 17.9
  Somewhat: Follow-up 4: number analyzed (Participants) | 136 | 124
  Somewhat: Follow-up 4 | 0 | 0
  Quite a bit: Follow-up 4: number analyzed (Participants) | 136 | 124
  Quite a bit: Follow-up 4 | 4.1 | 3.1
  Very much: Follow-up 4: number analyzed (Participants) | 136 | 124
  Very much: Follow-up 4 | 2.3 | 1.8

7. Secondary Outcome: Percentage of Participants by Response for Skin Problem Single Items
Description: Participants answered the Question 1 "Did itching skin bother you?" and Question 2 "Have you had skin problems?", from the mQLQ-BR23, on a 5-point scale (1 'Not at all', 2 'A little', 3 'Somewhat', 4 'Quite a bit', 5 'Very much'). Percentage of participants by each response was reported.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Number; unit: Percentage of Participants
Arm/Group | TCH + P | T-DM1 + P
Number analyzed (Participants) | 221 | 223
Percentage of Participants
  Q1: Not at all: Baseline: number analyzed (Participants) | 197 | 204
  Q1: Not at all: Baseline | 71.9 | 72.6
  Q1: A little bit: Baseline: number analyzed (Participants) | 197 | 204
  Q1: A little bit: Baseline | 14.9 | 16.1
  Q1: Somewhat: Baseline: number analyzed (Participants) | 197 | 204
  Q1: Somewhat: Baseline | 0 | 0
  Q1: Quite a bit: Baseline: number analyzed (Participants) | 197 | 204
  Q1: Quite a bit: Baseline | 2.3 | 2.2
  Q1: Very much: Baseline: number analyzed (Participants) | 197 | 204
  Q1: Very much: Baseline | 0 | 0.4
  Q1: Not at all: Neoadjuvant Cycle 3: number analyzed (Participants) | 176 | 183
  Q1: Not at all: Neoadjuvant Cycle 3 | 35.3 | 48.9
  Q1: A little bit: Neoadjuvant Cycle 3: number analyzed (Participants) | 176 | 183
  Q1: A little bit: Neoadjuvant Cycle 3 | 31.2 | 27.4
  Q1: Somewhat: Neoadjuvant Cycle 3: number analyzed (Participants) | 176 | 183
  Q1: Somewhat: Neoadjuvant Cycle 3 | 0 | 0
  Q1: Quite a bit: Neoadjuvant Cycle 3: number analyzed (Participants) | 176 | 183
  Q1: Quite a bit: Neoadjuvant Cycle 3 | 10.9 | 4.0
  Q1: Very much: Neoadjuvant Cycle 3: number analyzed (Participants) | 176 | 183
  Q1: Very much: Neoadjuvant Cycle 3 | 2.3 | 1.8
  Q1: Not at all: Neoadjuvant Cycle 5: number analyzed (Participants) | 181 | 178
  Q1: Not at all: Neoadjuvant Cycle 5 | 48.9 | 46.2
  Q1: A little bit: Neoadjuvant Cycle 5: number analyzed (Participants) | 181 | 178
  Q1: A little bit: Neoadjuvant Cycle 5 | 23.1 | 26.0
  Q1: Somewhat: Neoadjuvant Cycle 5: number analyzed (Participants) | 181 | 178
  Q1: Somewhat: Neoadjuvant Cycle 5 | 0 | 0
  Q1: Quite a bit: Neoadjuvant Cycle 5: number analyzed (Participants) | 181 | 178
  Q1: Quite a bit: Neoadjuvant Cycle 5 | 7.7 | 6.3
  Q1: Very much: Neoadjuvant Cycle 5: number analyzed (Participants) | 181 | 178
  Q1: Very much: Neoadjuvant Cycle 5 | 2.3 | 1.3
  Q1: Not at all: Pre-Surgery: number analyzed (Participants) | 170 | 171
  Q1: Not at all: Pre-Surgery | 40.3 | 48.0
  Q1: A little bit: Pre-Surgery: number analyzed (Participants) | 170 | 171
  Q1: A little bit: Pre-Surgery | 26.7 | 21.5
  Q1: Somewhat: Pre-Surgery: number analyzed (Participants) | 170 | 171
  Q1: Somewhat: Pre-Surgery | 0 | 0
  Q1: Quite a bit: Pre-Surgery: number analyzed (Participants) | 170 | 171
  Q1: Quite a bit: Pre-Surgery | 7.2 | 5.8
  Q1: Very much: Pre-Surgery: number analyzed (Participants) | 170 | 171
  Q1: Very much: Pre-Surgery | 2.7 | 1.3
  Q1: Not at all: Adjuvant Cycle 4: number analyzed (Participants) | 173 | 155
  Q1: Not at all: Adjuvant Cycle 4 | 38.5 | 39.0
  Q1: A little bit: Adjuvant Cycle 4: number analyzed (Participants) | 173 | 155
  Q1: A little bit: Adjuvant Cycle 4 | 23.5 | 21.5
  Q1: Somewhat: Adjuvant Cycle 4: number analyzed (Participants) | 173 | 155
  Q1: Somewhat: Adjuvant Cycle 4 | 0 | 0
  Q1: Quite a bit: Adjuvant Cycle 4: number analyzed (Participants) | 173 | 155
  Q1: Quite a bit: Adjuvant Cycle 4 | 9.5 | 6.7
  Q1: Very much: Adjuvant Cycle 4: number analyzed (Participants) | 173 | 155
  Q1: Very much: Adjuvant Cycle 4 | 6.8 | 2.2
  Q1: Not at all: Adjuvant Cycle 8: number analyzed (Participants) | 167 | 143
  Q1: Not at all: Adjuvant Cycle 8 | 34.8 | 39.0
  Q1: A little bit: Adjuvant Cycle 8: number analyzed (Participants) | 167 | 143
  Q1: A little bit: Adjuvant Cycle 8 | 27.6 | 15.7
  Q1: Somewhat: Adjuvant Cycle 8: number analyzed (Participants) | 167 | 143
  Q1: Somewhat: Adjuvant Cycle 8 | 0 | 0
  Q1: Quite a bit: Adjuvant Cycle 8: number analyzed (Participants) | 167 | 143
  Q1: Quite a bit: Adjuvant Cycle 8 | 9.0 | 6.3
  Q1: Very much: Adjuvant Cycle 8: number analyzed (Participants) | 167 | 143
  Q1: Very much: Adjuvant Cycle 8 | 4.1 | 3.1
  Q1: Not at all: End of Therapy: number analyzed (Participants) | 171 | 165
  Q1: Not at all: End of Therapy | 39.4 | 42.6
  Q1: A little bit: End of Therapy: number analyzed (Participants) | 171 | 165
  Q1: A little bit: End of Therapy | 26.7 | 22.9
  Q1: Somewhat: End of Therapy: number analyzed (Participants) | 171 | 165
  Q1: Somewhat: End of Therapy | 0 | 0
  Q1: Quite a bit: End of Therapy: number analyzed (Participants) | 171 | 165
  Q1: Quite a bit: End of Therapy | 6.8 | 6.7
  Q1: Very much: End of Therapy: number analyzed (Participants) | 171 | 165
  Q1: Very much: End of Therapy | 4.5 | 1.8
  Q1: Not at all: Follow-up 2: number analyzed (Participants) | 149 | 136
  Q1: Not at all: Follow-up 2 | 43.9 | 39.9
  Q1: A little bit: Follow-up 2: number analyzed (Participants) | 149 | 136
  Q1: A little bit: Follow-up 2 | 19.0 | 14.8
  Q1: Somewhat: Follow-up 2: number analyzed (Participants) | 149 | 136
  Q1: Somewhat: Follow-up 2 | 0 | 0
  Q1: Quite a bit: Follow-up 2: number analyzed (Participants) | 149 | 136
  Q1: Quite a bit: Follow-up 2 | 3.6 | 4.0
  Q1: Very much: Follow-up 2: number analyzed (Participants) | 149 | 136
  Q1: Very much: Follow-up 2 | 0.9 | 2.2
  Q1: Not at all: Follow-up 4: number analyzed (Participants) | 135 | 124
  Q1: Not at all: Follow-up 4 | 46.2 | 37.7
  Q1: A little bit: Follow-up 4: number analyzed (Participants) | 135 | 124
  Q1: A little bit: Follow-up 4 | 10.4 | 12.1
  Q1: Somewhat: Follow-up 4: number analyzed (Participants) | 135 | 124
  Q1: Somewhat: Follow-up 4 | 0 | 0
  Q1: Quite a bit: Follow-up 4: number analyzed (Participants) | 135 | 124
  Q1: Quite a bit: Follow-up 4 | 3.2 | 4.5
  Q1: Very much: Follow-up 4: number analyzed (Participants) | 135 | 124
  Q1: Very much: Follow-up 4 | 1.4 | 1.3
  Q2: Not at all: Baseline: number analyzed (Participants) | 198 | 204
  Q2: Not at all: Baseline | 64.7 | 67.3
  Q2: A little bit: Baseline: number analyzed (Participants) | 198 | 204
  Q2: A little bit: Baseline | 21.3 | 17.9
  Q2: Somewhat: Baseline: number analyzed (Participants) | 198 | 204
  Q2: Somewhat: Baseline | 0 | 0
  Q2: Quite a bit: Baseline: number analyzed (Participants) | 198 | 204
  Q2: Quite a bit: Baseline | 3.2 | 5.8
  Q2: Very much: Baseline: number analyzed (Participants) | 198 | 204
  Q2: Very much: Baseline | 0.5 | 0.4
  Q2: Not at all: Neoadjuvant Cycle 3: number analyzed (Participants) | 177 | 183
  Q2: Not at all: Neoadjuvant Cycle 3 | 14.0 | 24.2
  Q2: A little bit: Neoadjuvant Cycle 3: number analyzed (Participants) | 177 | 183
  Q2: A little bit: Neoadjuvant Cycle 3 | 40.7 | 38.6
  Q2: Somewhat: Neoadjuvant Cycle 3: number analyzed (Participants) | 177 | 183
  Q2: Somewhat: Neoadjuvant Cycle 3 | 0 | 0
  Q2: Quite a bit: Neoadjuvant Cycle 3: number analyzed (Participants) | 177 | 183
  Q2: Quite a bit: Neoadjuvant Cycle 3 | 18.6 | 14.8
  Q2: Very much: Neoadjuvant Cycle 3: number analyzed (Participants) | 177 | 183
  Q2: Very much: Neoadjuvant Cycle 3 | 6.8 | 4.5
  Q2: Not at all: Neoadjuvant Cycle 5: number analyzed (Participants) | 182 | 178
  Q2: Not at all: Neoadjuvant Cycle 5 | 21.3 | 25.6
  Q2: A little bit: Neoadjuvant Cycle 5: number analyzed (Participants) | 182 | 178
  Q2: A little bit: Neoadjuvant Cycle 5 | 35.7 | 37.7
  Q2: Somewhat: Neoadjuvant Cycle 5: number analyzed (Participants) | 182 | 178
  Q2: Somewhat: Neoadjuvant Cycle 5 | 0 | 0
  Q2: Quite a bit: Neoadjuvant Cycle 5: number analyzed (Participants) | 182 | 178
  Q2: Quite a bit: Neoadjuvant Cycle 5 | 20.4 | 12.6
  Q2: Very much: Neoadjuvant Cycle 5: number analyzed (Participants) | 182 | 178
  Q2: Very much: Neoadjuvant Cycle 5 | 5.0 | 4.0
  Q2: Not at all: Pre-Surgery: number analyzed (Participants) | 170 | 171
  Q2: Not at all: Pre-Surgery | 21.3 | 27.4
  Q2: A little bit: Pre-Surgery: number analyzed (Participants) | 170 | 171
  Q2: A little bit: Pre-Surgery | 33.9 | 37.2
  Q2: Somewhat: Pre-Surgery: number analyzed (Participants) | 170 | 171
  Q2: Somewhat: Pre-Surgery | 0 | 0
  Q2: Quite a bit: Pre-Surgery: number analyzed (Participants) | 170 | 171
  Q2: Quite a bit: Pre-Surgery | 15.4 | 8.1
  Q2: Very much: Pre-Surgery: number analyzed (Participants) | 170 | 171
  Q2: Very much: Pre-Surgery | 6.3 | 4.0
  Q2: Not at all: Adjuvant Cycle 4: number analyzed (Participants) | 174 | 155
  Q2: Not at all: Adjuvant Cycle 4 | 23.5 | 24.2
  Q2: A little bit: Adjuvant Cycle 4: number analyzed (Participants) | 174 | 155
  Q2: A little bit: Adjuvant Cycle 4 | 33.0 | 30.9
  Q2: Somewhat: Adjuvant Cycle 4: number analyzed (Participants) | 174 | 155
  Q2: Somewhat: Adjuvant Cycle 4 | 0 | 0
  Q2: Quite a bit: Adjuvant Cycle 4: number analyzed (Participants) | 174 | 155
  Q2: Quite a bit: Adjuvant Cycle 4 | 13.1 | 9.4
  Q2: Very much: Adjuvant Cycle 4: number analyzed (Participants) | 174 | 155
  Q2: Very much: Adjuvant Cycle 4 | 9.0 | 4.9
  Q2: Not at all: Adjuvant Cycle 8: number analyzed (Participants) | 168 | 143
  Q2: Not at all: Adjuvant Cycle 8 | 23.1 | 25.6
  Q2: A little bit: Adjuvant Cycle 8: number analyzed (Participants) | 168 | 143
  Q2: A little bit: Adjuvant Cycle 8 | 35.7 | 24.2
  Q2: Somewhat: Adjuvant Cycle 8: number analyzed (Participants) | 168 | 143
  Q2: Somewhat: Adjuvant Cycle 8 | 0 | 0
  Q2: Quite a bit: Adjuvant Cycle 8: number analyzed (Participants) | 168 | 143
  Q2: Quite a bit: Adjuvant Cycle 8 | 12.2 | 9.9
  Q2: Very much: Adjuvant Cycle 8: number analyzed (Participants) | 168 | 143
  Q2: Very much: Adjuvant Cycle 8 | 5.0 | 4.5
  Q2: Not at all: End of Therapy: number analyzed (Participants) | 172 | 165
  Q2: Not at all: End of Therapy | 27.1 | 27.4
  Q2: A little bit: End of Therapy: number analyzed (Participants) | 172 | 165
  Q2: A little bit: End of Therapy | 33.9 | 30.0
  Q2: Somewhat: End of Therapy: number analyzed (Participants) | 172 | 165
  Q2: Somewhat: End of Therapy | 0 | 0
  Q2: Quite a bit: End of Therapy: number analyzed (Participants) | 172 | 165
  Q2: Quite a bit: End of Therapy | 10.0 | 13.5
  Q2: Very much: End of Therapy: number analyzed (Participants) | 172 | 165
  Q2: Very much: End of Therapy | 6.8 | 3.1
  Q2: Not at all: Follow-up 2: number analyzed (Participants) | 150 | 136
  Q2: Not at all: Follow-up 2 | 36.2 | 27.8
  Q2: A little bit: Follow-up 2: number analyzed (Participants) | 150 | 136
  Q2: A little bit: Follow-up 2 | 25.8 | 25.6
  Q2: Somewhat: Follow-up 2: number analyzed (Participants) | 150 | 136
  Q2: Somewhat: Follow-up 2 | 0 | 0
  Q2: Quite a bit: Follow-up 2: number analyzed (Participants) | 150 | 136
  Q2: Quite a bit: Follow-up 2 | 4.1 | 6.3
  Q2: Very much: Follow-up 2: number analyzed (Participants) | 150 | 136
  Q2: Very much: Follow-up 2 | 1.8 | 1.3
  Q2: Not at all: Follow-up 4: number analyzed (Participants) | 136 | 124
  Q2: Not at all: Follow-up 4 | 39.8 | 30.0
  Q2: A little bit: Follow-up 4: number analyzed (Participants) | 136 | 124
  Q2: A little bit: Follow-up 4 | 14.5 | 18.8
  Q2: Somewhat: Follow-up 4: number analyzed (Participants) | 136 | 124
  Q2: Somewhat: Follow-up 4 | 0 | 0
  Q2: Quite a bit: Follow-up 4: number analyzed (Participants) | 136 | 124
  Q2: Quite a bit: Follow-up 4 | 4.5 | 4.5
  Q2: Very much: Follow-up 4: number analyzed (Participants) | 136 | 124
  Q2: Very much: Follow-up 4 | 2.7 | 2.2

8. Secondary Outcome: Percentage of Participants With a Clinically Meaningful Deterioration in Global Health Status (GHS)/Quality of Life (QoL) Score
Description: Participants rated their quality of life (global health status) on European Organization for the Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ- C30), with total scores ranging from 0 (worst) to 100 (best); where higher score indicates better quality of life. Clinically meaningful deterioration in GHS/QoL was defined as a decrease in score of 10 points in GHS/QoL.
Time Frame: From Baseline (Day 1 Cycle 1) to Cycle 6 (each cycle = 21 days) in neoadjuvant period
Population: The Intent-to-treat (ITT) Population comprised all randomized participants, whether or not they received any study treatment or completed a full course of study treatment. Participants were analyzed according to their randomized treatment. As per protocol, the analysis for this outcome measure was focused on the neoadjuvant period only.
Measure: Number; unit: Percentage of Participants
Arm/Group | TCH + P | T-DM1 + P
Number analyzed (Participants) | 193 | 205
Percentage of Participants | 69.9 | 45.4
Statistical Analysis 1: Comparison: TCH + P vs T-DM1 + P; 95% CI for the difference in clinically meaningful deterioration in GHS/QoL score between treatment arms was calculated using normal approximation; Test type: Superiority; Difference in Deterioration = -24.58, 95% CI 2-sided [-33.98 to -15.19]

9. Secondary Outcome: Time to Clinically Meaningful Deterioration in GHS/QoL Score
Description: Participants rated their quality of life (global health status) on EORTC QLQ C-30, with total scores ranging from 0 (worst) to 100 (best); where higher score indicates better quality of life. Time to deterioration was defined as the time from baseline to first 10-point (or greater) decrease as measured by GHS/QoL. All valid GHS/QoL questionnaires of the neoadjuvant phase including surgery were used. Participants without deterioration were censored at the time of completing the last GHS/QoL plus 1 day. Median time to deterioration was estimated with Kaplan-Meier method. The 95% confidence interval (CI) for the median was computed using the method of Brookmeyer and Crowley.
Time Frame: From Baseline (Day 1 Cycle 1) to Cycle 6 (each cycle = 21 days) in neoadjuvant period
Population: as for outcome 8
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TCH + P | T-DM1 + P
Number analyzed (Participants) | 191 | 200
months | 3.02 (2.83) [2.83 to 3.38] | 4.63 (4.11) [4.11 to 7.98]
Statistical Analysis 1: Comparison: TCH + P vs T-DM1 + P; Stratified cox proportional hazards regression model was used to estimate Hazard Ratio and CI. Stratification by hormonal receptor status and clinical stage at presentation (stratification factors); Test type: Superiority; p = 0.0001, Log Rank; Log Rank was used and stratified by local hormone receptor status and clinical stage at presentation; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.46 to 0.78]

10. Secondary Outcome: Time to Clinically Meaningful Deterioration in Function Subscale
Description: Participants rated their function on EORTC QLQ C-30, with total scores ranging from 0 (worst) to 100 (best); where higher score indicates better functioning. Time to deterioration was defined as the time from baseline to first 10-point (or greater) decrease as measured by physical function; to first 14-point (or greater) decrease as measured by role function, to first 7-point (or greater) decrease as measured by cognitive function. Median time to deterioration was estimated with Kaplan-Meier method. The 95% CI for the median was computed using the method of Brookmeyer and Crowley.
Time Frame: From Baseline (Day 1 Cycle 1) to Cycle 6 (each cycle = 21 days) in neoadjuvant period
Population: Patients of the ITT population with a baseline assessment and at least one post-treatment assessment was included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TCH + P | T-DM1 + P
Number analyzed (Participants) | 191 | 200
months
  Physical Function | 2.79 [2.79 to 2.96] | 4.86 [4.40 to 7.98]
  Role Function | 2.79 [2.17 to 2.89] | 4.44 [4.04 to 4.53]
  Cognitive Function | 3.42 [3.02 to 4.24] | 4.44 [4.21 to NA] — Upper limit not reached.

11. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of Trastuzumab
Description: Only participants who received trastuzumab were to be analyzed for this outcome.
Time Frame: 15-30 minutes (min) post-study treatment infusion (infusion duration = 90 min) on Day 1 of Cycle 1 and 6 (each cycle = 21 days) in neoadjuvant and adjuvant period
Population: The pharmacokinetic population comprised all patients who received at least one treatment dose of trastuzumab emtansine (for patients in the T-DM1 + P arm) or trastuzumab (for patients in the TCH + P arm), and had at least one post-treatment serum or plasma sample.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | TCH + P
Number analyzed (Participants) | 214
micrograms per milliliter (mcg/mL)
  Cycle 1 (neoadjuvant period): number analyzed (Participants) | 162
  Cycle 1 (neoadjuvant period) | 167 (47.1)
  Cycle 6 (neoadjuvant period): number analyzed (Participants) | 155
  Cycle 6 (neoadjuvant period) | 148 (44.7)
  Cycle 1 (adjuvant period): number analyzed (Participants) | 97
  Cycle 1 (adjuvant period) | 159 (36.2)
  Cycle 6 (adjuvant period): number analyzed (Participants) | 49
  Cycle 6 (adjuvant period) | 181 (30.7)

12. Secondary Outcome: Cmax of Trastuzumab Emtansine and Total Trastuzumab
Description: Only participants who received trastuzumab emtansine were to be analyzed for this outcome.
Time Frame: 15-30 min post-study treatment infusion (infusion duration = 90 min) on Day 1 of Cycle 1 and 6 (each cycle = 21 days) in neoadjuvant and adjuvant period.
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | T-DM1 + P
Number analyzed (Participants) | 222
mcg/mL
  Trastuzumab emtansine: C1 (neoadjuvant): number analyzed (Participants) | 207
  Trastuzumab emtansine: C1 (neoadjuvant) | 80.4 (26.5)
  Trastuzumab emtansine: C6 (neoadjuvant): number analyzed (Participants) | 190
  Trastuzumab emtansine: C6 (neoadjuvant) | 71.7 (30.2)
  Total Trastuzumab: C1 (neoadjuvant): number analyzed (Participants) | 208
  Total Trastuzumab: C1 (neoadjuvant) | 79.1 (25.7)
  Total Trastuzumab: C6 (neoadjuvant): number analyzed (Participants) | 190
  Total Trastuzumab: C6 (neoadjuvant) | 79.1 (31.1)
  Trastuzumab emtansine: C1 (adjuvant): number analyzed (Participants) | 165
  Trastuzumab emtansine: C1 (adjuvant) | 70.4 (22.7)
  Trastuzumab emtansine: C6 (adjuvant): number analyzed (Participants) | 141
  Trastuzumab emtansine: C6 (adjuvant) | 73.1 (21.8)
  Total Trastuzumab: C1 (adjuvant): number analyzed (Participants) | 165
  Total Trastuzumab: C1 (adjuvant) | 73.0 (23.2)
  Total Trastuzumab: C6 (adjuvant): number analyzed (Participants) | 141
  Total Trastuzumab: C6 (adjuvant) | 82.6 (23.7)

13. Secondary Outcome: Minimum Observed Serum Concentration (Cmin) of Trastuzumab
Description: Only participants who received trastuzumab were to be analyzed for this outcome.
Time Frame: Pre-study treatment infusion (0 hours [hr]) (infusion duration = 90 min) on Day 1 of Cycle 6 (cycle length = 21 days) in neoadjuvant and adjuvant period
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | TCH + P
Number analyzed (Participants) | 214
mcg/mL
  Trastuzumab (neoadjuvant period): number analyzed (Participants) | 165
  Trastuzumab (neoadjuvant period) | 45.8 (17.8)
  Trastuzumab (adjuvant period): number analyzed (Participants) | 3
  Trastuzumab (adjuvant period) | 21.8 (0.153)

14. Secondary Outcome: Cmin of Trastuzumab Emtansine and Total Trastuzumab
Description: Only participants who received trastuzumab emtansine were to be analyzed for this outcome.
Time Frame: Pre-study treatment infusion (0 hr) (infusion duration = 90 min) on Day 1 of Cycle 6 (cycle length = 21 days) in neoadjuvant and adjuvant period
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | T-DM1 + P
Number analyzed (Participants) | 222
mcg/mL
  Trastuzumab emtansine (neoadjuvant): number analyzed (Participants) | 203
  Trastuzumab emtansine (neoadjuvant) | 3.04 (7.43)
  Total Trastuzumab (neoadjuvant): number analyzed (Participants) | 204
  Total Trastuzumab (neoadjuvant) | 12.3 (8.68)
  Trastuzumab emtansine (adjuvant): number analyzed (Participants) | 149
  Trastuzumab emtansine (adjuvant) | 4.09 (11.7)
  Total Trastuzumab (adjuvant): number analyzed (Participants) | 149
  Total Trastuzumab (adjuvant) | 8.70 (6.98)

15. Secondary Outcome: Plasma N2'-Deacetyl-N2'-(3-mercapto-1-oxopropyl)-Maytansine (DM1) Concentrations
Description: DM1 is the metabolite of trastuzumab emtansine. Only participants who received trastuzumab emtansine were to be analyzed for this outcome.
Time Frame: 15-30 min post-study treatment infusion (Cmax) on Day 1 of Cycle 1 and 6 in neoadjuvant and adjuvant period
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | T-DM1 + P
Number analyzed (Participants) | 222
nanograms per milliliter (ng/mL)
  C1: 15-30 min post-dose (neoadjuvant): number analyzed (Participants) | 173
  C1: 15-30 min post-dose (neoadjuvant) | 4.64 (2.33)
  C6: 15-30 min post-dose (neoadjuvant): number analyzed (Participants) | 163
  C6: 15-30 min post-dose (neoadjuvant) | 4.73 (2.61)
  C1: 15-30 min post-dose (adjuvant): number analyzed (Participants) | 146
  C1: 15-30 min post-dose (adjuvant) | 4.49 (2.33)
  C6: 15-30 min post-dose (adjuvant): number analyzed (Participants) | 119
  C6: 15-30 min post-dose (adjuvant) | 5.15 (8.28)

16. Secondary Outcome: Serum Levels of Plasma DM1-Containing Catabolites Concentrations (in ng/mL) (Nonreducible Thioether Linker [MCC]-DM1 and Lysine [Lys]-MCC-DM1)
Time Frame: 15-30 min post-study treatment infusion (Cmax) on Day 1 of Cycle 1 and 6 in neoadjuvant and adjuvant period
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | T-DM1 + P
Number analyzed (Participants) | 222
ng/mL
  C1: MCC-DM1 (Neoadjuvant Period): number analyzed (Participants) | 131
  C1: MCC-DM1 (Neoadjuvant Period) | 8.18 (7.23)
  C1: Lys-MCC-DM1 (Neoadjuvant period) | NA (NA) — not reported since more than 1/3 of the results are LTR (Lower than reportable)
  C6: MCC-DM1 (Neoadjuvant Period): number analyzed (Participants) | 100
  C6: MCC-DM1 (Neoadjuvant Period) | 8.22 (8.03)
  C6: Lys-MCC-DM1 (Neoadjuvant period) | NA (NA) — not reported since more than 1/3 of the results are LTR (Lower than reportable)
  C1: MCC-DM1 (Adjuvant Period): number analyzed (Participants) | 96
  C1: MCC-DM1 (Adjuvant Period) | 7.98 (6.46)
  C1: Lys-MCC-DM1 (Adjuvant period) | NA (NA) — not reported since more than 1/3 of the results are LTR (Lower than reportable)
  C6: MCC-DM1 (Adjuvant Period): number analyzed (Participants) | 76
  C6: MCC-DM1 (Adjuvant Period) | 7.90 (5.37)
  C6: Lys-MCC-DM1 (Adjuvant period) | NA (NA) — not reported since more than 1/3 of the results are LTR (Lower than reportable)

17. Secondary Outcome: Percentage of Participants With ATA to Trastuzumab
Time Frame: Baseline (Pre-trastuzumab [0 hr] infusion [infusion duration = 90 min] on Day 1 of Cycle 1); post-baseline (Pre-trastuzumab infusion [0 hr] on Day 1 of Cycle 6) (each cycle = 21 days) in neoadjuvant and adjuvant period
Population: The participants included in this analysis were the participants who received at least one dose of trastuzumab and had at least one reported serum or plasma results.
Measure: Number; unit: Percentage of participants
Arm/Group | T-DM1 + P
Number analyzed (Participants) | 210
Percentage of participants
  Neoadjuvant Phase (baseline) | 11
  Neoadjuvant Phase (post-baseline): number analyzed (Participants) | 191
  Neoadjuvant Phase (post-baseline) | 2.6
  Adjuvant Phase (baseline): number analyzed (Participants) | 129
  Adjuvant Phase (baseline) | 5.4
  Adjuvant Phase (post-baseline): number analyzed (Participants) | 60
  Adjuvant Phase (post-baseline) | 5.0

18. Secondary Outcome: Percentage of Participants by Response for Hair Loss Single Item
Description: Participants answered the Question "Have you lost any hair?", from the mQLQ-BR23, on a 5-point scale (1 'Not at all', 2 'A little', 3 'Somewhat', 4 'Quite a bit', 5 'Very much'). Percentage of participants by each response was reported.
Time Frame: Baseline,Cycle(C) 3, C5 of neoadjuvant period (each C=21 days); pre-surgery visit (within 6weeks after neoadjuvant therapy; up to approx 6months), C4 & 8 of Adjuvant Period (each C=21 days), End of Treatment, Follow up 2 & 4(approx 47 months)
Population: as for outcome 6
Measure: Number; unit: Percentage of Participants
Arm/Group | TCH + P | T-DM1 + P
Number analyzed (Participants) | 221 | 223
Percentage of Participants
  Not at all: Baseline: number analyzed (Participants) | 198 | 204
  Not at all: Baseline | 81.4 | 87.4
  A little bit: Baseline: number analyzed (Participants) | 198 | 204
  A little bit: Baseline | 7.7 | 4.0
  Somewhat: Baseline: number analyzed (Participants) | 198 | 204
  Somewhat: Baseline | 0 | 0
  Quite a bit: Baseline: number analyzed (Participants) | 198 | 204
  Quite a bit: Baseline | 0.5 | 0
  Very much: Baseline: number analyzed (Participants) | 198 | 204
  Very much: Baseline | 0 | 0
  Not at all: Neoadjuvant Cycle 3: number analyzed (Participants) | 177 | 183
  Not at all: Neoadjuvant Cycle 3 | 8.6 | 65.0
  A little bit: Neoadjuvant Cycle 3: number analyzed (Participants) | 177 | 183
  A little bit: Neoadjuvant Cycle 3 | 11.3 | 16.6
  Somewhat: Neoadjuvant Cycle 3: number analyzed (Participants) | 177 | 183
  Somewhat: Neoadjuvant Cycle 3 | 0 | 0
  Quite a bit: Neoadjuvant Cycle 3: number analyzed (Participants) | 177 | 183
  Quite a bit: Neoadjuvant Cycle 3 | 20.8 | 0.4
  Very much: Neoadjuvant Cycle 3: number analyzed (Participants) | 177 | 183
  Very much: Neoadjuvant Cycle 3 | 39.4 | 0
  Not at all: Neoadjuvant Cycle 5: number analyzed (Participants) | 182 | 178
  Not at all: Neoadjuvant Cycle 5 | 20.4 | 58.7
  A little bit: Neoadjuvant Cycle 5: number analyzed (Participants) | 182 | 178
  A little bit: Neoadjuvant Cycle 5 | 19.9 | 19.3
  Somewhat: Neoadjuvant Cycle 5: number analyzed (Participants) | 182 | 178
  Somewhat: Neoadjuvant Cycle 5 | 0 | 0
  Quite a bit: Neoadjuvant Cycle 5: number analyzed (Participants) | 182 | 178
  Quite a bit: Neoadjuvant Cycle 5 | 15.8 | 1.3
  Very much: Neoadjuvant Cycle 5: number analyzed (Participants) | 182 | 178
  Very much: Neoadjuvant Cycle 5 | 26.2 | 0.4
  Not at all: Pre-Surgery: number analyzed (Participants) | 170 | 171
  Not at all: Pre-Surgery | 30.8 | 49.8
  A little bit: Pre-Surgery: number analyzed (Participants) | 170 | 171
  A little bit: Pre-Surgery | 13.6 | 24.7
  Somewhat: Pre-Surgery: number analyzed (Participants) | 170 | 171
  Somewhat: Pre-Surgery | 0 | 0
  Quite a bit: Pre-Surgery: number analyzed (Participants) | 170 | 171
  Quite a bit: Pre-Surgery | 11.3 | 2.2
  Very much: Pre-Surgery: number analyzed (Participants) | 170 | 171
  Very much: Pre-Surgery | 21.3 | 0
  Not at all: Adjuvant Cycle 4: number analyzed (Participants) | 174 | 155
  Not at all: Adjuvant Cycle 4 | 67.9 | 50.2
  A little bit: Adjuvant Cycle 4: number analyzed (Participants) | 174 | 155
  A little bit: Adjuvant Cycle 4 | 5.0 | 15.7
  Somewhat: Adjuvant Cycle 4: number analyzed (Participants) | 174 | 155
  Somewhat: Adjuvant Cycle 4 | 0 | 0
  Quite a bit: Adjuvant Cycle 4: number analyzed (Participants) | 174 | 155
  Quite a bit: Adjuvant Cycle 4 | 3.2 | 2.2
  Very much: Adjuvant Cycle 4: number analyzed (Participants) | 174 | 155
  Very much: Adjuvant Cycle 4 | 2.7 | 1.3
  Not at all: Adjuvant Cycle 8: number analyzed (Participants) | 168 | 143
  Not at all: Adjuvant Cycle 8 | 70.1 | 48.9
  A little bit: Adjuvant Cycle 8: number analyzed (Participants) | 168 | 143
  A little bit: Adjuvant Cycle 8 | 4.1 | 14.3
  Somewhat: Adjuvant Cycle 8: number analyzed (Participants) | 168 | 143
  Somewhat: Adjuvant Cycle 8 | 0 | 0
  Quite a bit: Adjuvant Cycle 8: number analyzed (Participants) | 168 | 143
  Quite a bit: Adjuvant Cycle 8 | 0.9 | 0.9
  Very much: Adjuvant Cycle 8: number analyzed (Participants) | 168 | 143
  Very much: Adjuvant Cycle 8 | 0.9 | 0
  Not at all: End of Therapy: number analyzed (Participants) | 172 | 165
  Not at all: End of Therapy | 69.7 | 57.8
  A little bit: End of Therapy: number analyzed (Participants) | 172 | 165
  A little bit: End of Therapy | 5.4 | 14.8
  Somewhat: End of Therapy: number analyzed (Participants) | 172 | 165
  Somewhat: End of Therapy | 0 | 0
  Quite a bit: End of Therapy: number analyzed (Participants) | 172 | 165
  Quite a bit: End of Therapy | 0.9 | 0
  Very much: End of Therapy: number analyzed (Participants) | 172 | 165
  Very much: End of Therapy | 1.8 | 1.3
  Not at all: Follow-up 2: number analyzed (Participants) | 150 | 136
  Not at all: Follow-up 2 | 55.7 | 48.4
  A little bit: Follow-up 2: number analyzed (Participants) | 150 | 136
  A little bit: Follow-up 2 | 9.0 | 11.7
  Somewhat: Follow-up 2: number analyzed (Participants) | 150 | 136
  Somewhat: Follow-up 2 | 0 | 0
  Quite a bit: Follow-up 2: number analyzed (Participants) | 150 | 136
  Quite a bit: Follow-up 2 | 1.4 | 0.4
  Very much: Follow-up 2: number analyzed (Participants) | 150 | 136
  Very much: Follow-up 2 | 1.8 | 0.4
  Not at all: Follow-up 4: number analyzed (Participants) | 136 | 124
  Not at all: Follow-up 4 | 52.9 | 41.3
  A little bit: Follow-up 4: number analyzed (Participants) | 136 | 124
  A little bit: Follow-up 4 | 7.2 | 11.2
  Somewhat: Follow-up 4: number analyzed (Participants) | 136 | 124
  Somewhat: Follow-up 4 | 0 | 0
  Quite a bit: Follow-up 4: number analyzed (Participants) | 136 | 124
  Quite a bit: Follow-up 4 | 0 | 2.7
  Very much: Follow-up 4: number analyzed (Participants) | 136 | 124
  Very much: Follow-up 4 | 1.4 | 0.4

19. Secondary Outcome: Percentage of Participants With Selected Adverse Events (AEs)
Description: Selected AEs included hepatotoxicity, pulmonary toxicity, cardiac dysfunction, neutropenia, thrombocytopenia, peripheral neuropathy, hemorrhage, infusion related reaction (IRR)/hypersensitivity, IRR/Hypersensitivity symptoms, rash, diarrhea and mucositis. An AE was defined as any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product, regardless of causal attribution.
Time Frame: Baseline to end of study (approximately 47 months)
Population: The Safety Population comprised all patients who received at least one full or partial dose of any study treatment. Patients were analyzed according to the treatment they actually received.
Measure: Number; unit: Percentage of Participants
Arm/Group | TCH + P | T-DM1 + P
Number analyzed (Participants) | 219 | 223
Percentage of Participants
  Hepatotoxicity | 14.2 | 39.0
  Pulmonary Toxicity | 0.9 | 4.9
  Cardiac Dysfunction | 4.6 | 1.3
  Neutropenia | 39.7 | 8.1
  Thrombocytopenia | 22.8 | 17.9
  Peripheral Neuropathy | 47.5 | 28.7
  Hemorrhage | 19.2 | 33.2
  IRR/Hypersensitivity | 13.7 | 22.9
  IRR/Hypersensitivity symptoms | 7.8 | 19.3
  Rash | 44.7 | 36.8
  Diarrhea | 76.7 | 38.6
  Mucositis | 43.8 | 24.7

20. Secondary Outcome: Percentage of Participants With a Clinically Meaningful Deterioration in Function Subscales
Description: Participants rated their function on EORTC QLQ C-30, with total score and single-item (physical, cognitive and role functioning) scores ranging from 0 (worst) to 100 (best); where higher score indicates better functioning. Clinically meaningful deterioration was defined as a decrease in score of 10 points in physical function; decrease of 7 points in cognitive function and decrease of 14 points in role function.
Time Frame: From Baseline (Day 1 Cycle 1) to Cycle 6 (each cycle = 21 days) in neoadjuvant period
Population: as for outcome 8
Measure: Number; unit: Percentage of Participants
Arm/Group | TCH + P | T-DM1 + P
Number analyzed (Participants) | 193 | 205
Percentage of Participants
  Cognitive Functioning | 59.1 | 42.4
  Physical Functioning | 72.5 | 40.0
  Role Functioning | 76.7 | 47.8
Statistical Analysis 1: Comparison: TCH + P vs T-DM1 + P; This is the statistical analysis for cognitive functioning. 95% CI for the difference in clinically meaningful deterioration in function subscales between treatment arms was calculated using normal approximation; Test type: Superiority; Difference in Deterioration = -16.63, 95% CI 2-sided [-26.32 to -6.94]
Statistical Analysis 2: Comparison: TCH + P vs T-DM1 + P; This is the statistical analysis for physical functioning. 95% CI for the difference in clinically meaningful deterioration in function subscales between treatment arms was calculated using normal approximation; Test type: Superiority; Difference in Deterioration = -32.54, 95% CI 2-sided [-41.74 to -23.34]
Statistical Analysis 3: Comparison: TCH + P vs T-DM1 + P; This is the statistical analysis for role functioning. 95% CI for the difference in clinically meaningful deterioration in function subscales between treatment arms was calculated using normal approximation; Test type: Superiority; Difference in Deterioration = -28.88, 95% CI 2-sided [-37.95 to -19.80]

21. Secondary Outcome: Percentage of Participants With Anti-Therapeutic Antibodies (ATA) to TDM-1
Description: Participants were considered post-baseline ATA positive if they had ATAs post-baseline that were either treatment-induced or treatment-enhanced. Participants had treatment-induced ATAs if they had a negative or missing ATA result at baseline, and at least one positive ATA result post-baseline. Participants had treatment-enhanced ATAs if they had a positive ATA result at baseline, and at least one positive ATA result post-baseline that was greater than or equal to (>/=) 0.60 titer units higher than the result at baseline.
Time Frame: Baseline (b) (Pre-TDM1 [0 hr] infusion [infusion duration = 90 min] on Day 1 of Cycle 1); post-baseline (pb) (Pre-TDM1 infusion [0 hr] on Day 1 of Cycle 6) (each cycle = 21 days) in neoadjuvant and adjuvant period
Population: The participants included in this analysis were the participants who received at least one dose of trastuzumab emtansine and had at least one reported serum or plasma results.
Measure: Number; unit: Percentage of Participants
Arm/Group | T-DM1 + P
Number analyzed (Participants) | 219
Percentage of Participants
  Neoadjuvant Phase (Baseline) | 5.5
  Neoadjuvant Phase (Post-Baseline): number analyzed (Participants) | 214
  Neoadjuvant Phase (Post-Baseline) | 7.5
  Adjuvant Phase (Baseline): number analyzed (Participants) | 180
  Adjuvant Phase (Baseline) | 11.7
  Adjuvant Phase (Post-baseline): number analyzed (Participants) | 191
  Adjuvant Phase (Post-baseline) | 13.1

22. Secondary Outcome: Percentage of Participants With a Clinically Meaningful Increase in Symptom Subscales
Description: Participants rated their symptoms on EORTC QLQ C-30 and mQLQ-BR23, with total scores ranging from 0 (worst) to 100 (best); where higher score indicates greater degree of symptoms. Clinically meaningful increase in symptoms was defined as an increase in score (deterioration) of 11 points in nausea and vomiting, pain, dyspnea; increase of 9 points in insomnia; increase of 14 points in appetite loss; increase of 15 points in diarrhea, constipation; increase of 10 points in fatigue, systemic therapy side effects, hair loss.
Time Frame: From Baseline (Day 1 Cycle 1) to Cycle 6 (each cycle = 21 days) in neoadjuvant period
Population: as for outcome 8
Measure: Number; unit: Percentage of Participants
Arm/Group | TCH + P | T-DM1 + P
Number analyzed (Participants) | 194 | 205
Percentage of Participants
  Appetite Loss | 61.1 | 47.8
  Any Hair Loss | 91.2 | 40.5
  Systemic Therapy Side-Effects | 89.7 | 75.1
  Constipation | 33.2 | 32.7
  Diarrhea | 79.3 | 50.7
  Dyspnea | 56.0 | 31.2
  Fatigue | 87.6 | 68.8
  Nausea/Vomiting | 66.3 | 43.9
  Pain | 56.0 | 36.6
  Insomnia | 42.5 | 30.2

ADVERSE EVENTS:
Time Frame: From Baseline up to approximately 47 months
Description: Safety population was analyzed.
Arm/Group | TCH + P | T-DM1 + P
All-Cause Mortality (participants affected / at risk) | 5/219 | 6/223
Serious Adverse Events (participants affected / at risk) | 70/219 | 30/223
Other Adverse Events (participants affected / at risk) | 217/219 | 212/223
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | TCH + P (N=219) | T-DM1 + P (N=223)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 26 (33) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 7 (7) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 2 (2) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 3 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 9 (9) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Breast cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (2) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis norovirus (Infections and infestations) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 2 (2)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 3 (3)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 3 (3) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Adenomyosis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast haematoma (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0)
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Device related thrombosis (General disorders) | 1 (1) | 0 (0)
Nodular regenerative hyperplasia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Breast abscess (Infections and infestations) | 0 (0) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cervix carinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0/0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TCH + P (N=219) | T-DM1 + P (N=223)
Anaemia (Blood and lymphatic system disorders) | 81 (103) | 43 (47)
Neutropenia (Blood and lymphatic system disorders) | 59 (92) | 13 (20)
Thrombocytopenia (Blood and lymphatic system disorders) | 24 (36) | 18 (23)
Dry eye (Eye disorders) | 14 (16) | 16 (16)
Lacrimation increased (Eye disorders) | 18 (21) | 6 (9)
Abdominal pain (Gastrointestinal disorders) | 30 (45) | 21 (29)
Abdominal pain upper (Gastrointestinal disorders) | 22 (29) | 7 (8)
Constipation (Gastrointestinal disorders) | 43 (48) | 34 (52)
Diarrhoea (Gastrointestinal disorders) | 163 (372) | 86 (179)
Dry mouth (Gastrointestinal disorders) | 4 (4) | 27 (33)
Dyspepsia (Gastrointestinal disorders) | 15 (18) | 25 (30)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 16 (18) | 7 (8)
Haemorrhoids (Gastrointestinal disorders) | 14 (19) | 5 (5)
Nausea (Gastrointestinal disorders) | 139 (249) | 103 (248)
Stomatitis (Gastrointestinal disorders) | 49 (70) | 23 (30)
Vomiting (Gastrointestinal disorders) | 68 (83) | 35 (47)
Asthenia (General disorders) | 61 (115) | 42 (73)
Chills (General disorders) | 9 (9) | 27 (32)
Fatigue (General disorders) | 95 (143) | 83 (116)
Influenza like illness (General disorders) | 10 (12) | 16 (21)
Mucosal inflammation (General disorders) | 30 (37) | 22 (29)
Oedema peripheral (General disorders) | 31 (38) | 10 (11)
Pyrexia (General disorders) | 34 (43) | 38 (53)
Nasopharyngitis (Infections and infestations) | 23 (29) | 29 (34)
Upper respiratory tract infection (Infections and infestations) | 15 (18) | 21 (24)
Urinary tract infection (Infections and infestations) | 17 (20) | 12 (16)
Radiation skin injury (Injury, poisoning and procedural complications) | 46 (48) | 21 (22)
Alanine aminotransferase increased (Investigations) | 24 (37) | 64 (83)
Aspartate aminotransferase increased (Investigations) | 21 (37) | 55 (74)
Neutrophil count decreased (Investigations) | 22 (44) | 5 (6)
Platelet count decreased (Investigations) | 26 (37) | 23 (38)
Weight decreased (Investigations) | 24 (24) | 18 (19)
White blood cell count decreased (Investigations) | 17 (22) | 8 (11)
Decreased appetite (Metabolism and nutrition disorders) | 40 (46) | 33 (41)
Hypokalaemia (Metabolism and nutrition disorders) | 20 (23) | 13 (17)
Hypomagnesaemia (Metabolism and nutrition disorders) | 13 (13) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 41 (55) | 31 (37)
Back pain (Musculoskeletal and connective tissue disorders) | 20 (22) | 14 (20)
Bone pain (Musculoskeletal and connective tissue disorders) | 17 (25) | 8 (8)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 14 (16) | 20 (21)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 20 (22) | 10 (10)
Myalgia (Musculoskeletal and connective tissue disorders) | 37 (41) | 28 (42)
Dizziness (Nervous system disorders) | 27 (30) | 22 (28)
Dysgeusia (Nervous system disorders) | 44 (58) | 31 (39)
Headache (Nervous system disorders) | 37 (53) | 68 (95)
Hypoaesthesia (Nervous system disorders) | 19 (21) | 7 (9)
Neuropathy peripheral (Nervous system disorders) | 29 (36) | 21 (37)
Paraesthesia (Nervous system disorders) | 23 (28) | 11 (14)
Peripheral sensory neuropathy (Nervous system disorders) | 26 (26) | 26 (27)
Depression (Psychiatric disorders) | 16 (17) | 10 (10)
Insomnia (Psychiatric disorders) | 31 (37) | 36 (40)
Breast pain (Reproductive system and breast disorders) | 12 (13) | 17 (18)
Cough (Respiratory, thoracic and mediastinal disorders) | 21 (26) | 30 (38)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18 (21) | 18 (22)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 24 (31) | 49 (82)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 11 (17) | 10 (11)
Alopecia (Skin and subcutaneous tissue disorders) | 146 (149) | 37 (38)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 16 (16) | 12 (14)
Dry skin (Skin and subcutaneous tissue disorders) | 27 (32) | 30 (32)
Nail discolouration (Skin and subcutaneous tissue disorders) | 20 (21) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 11 (13) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 26 (34) | 20 (22)
Rash (Skin and subcutaneous tissue disorders) | 57 (77) | 43 (60)
Hot flush (Vascular disorders) | 45 (47) | 22 (25)
Hypertension (Vascular disorders) | 15 (18) | 14 (14)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 15 (17)
Hypersensitivity (Immune system disorders) | 11 (17) | 6 (8)
Blood bilirubin increased (Investigations) | 1 (3) | 20 (28)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 (16) | 15 (15)
Anxiety (Psychiatric disorders) | 14 (15) | 13 (15)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 12 (16) | 11 (14)
Erythema (Skin and subcutaneous tissue disorders) | 8 (10) | 16 (18)

LIMITATIONS AND CAVEATS:
The reported results are interim only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.